CLINICAL TRIAL: NCT03327883
Title: Retrospective Review of FDG PET MRI Management of Patients With Muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918009; 18-C-N009
Record Dates: First submitted 2017-10-31; First posted 2017-11-01 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
Keywords: Diagnostic Imaging; Review of Patients Records; PET MRI; Treatment Responses
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- 1/Patients medical records: Medical records of patients with metastatic bladder cancer

SUMMARY:
Background:

Bladder cancer is a common cancer in the U.S. Survival rates for metastatic bladder cancer have not gotten better for 15 years. Diagnosing and assessing the disease is important for treating it. The best way to tell what stage a cancer is in is computed tomography. This is also called CT. But it does not always give the best images of the bladder. Adding a test called positron emission tomography (PET) can help. Magnetic resonance imaging (MRI) is even better than CT for detecting bladder cancer. But it is not widely used.

Some people with bladder cancer have already had MRI/PET and CT. Researchers want to study their records. They want to compare the different ways of assessing the disease.

Objective:

To evaluate the use of MRI/PET for diagnosing and treating metastatic bladder cancer.

Eligibility:

People 18 years and older who were in studies between 2013 and 2016

Design:

Researchers will study existing records. There will be no active participants.

The records will have no data that could identify the participants. Data will be stored on secure computers.

No study participants will be contacted without approval from a review board.

DETAILED DESCRIPTION:
This protocol is a chart review of the diagnostic imaging and management of patients with metastatic bladder cancer who have undergone PET MRI. The study will involve only review of patient records and will not use specimens or participant contact. The participants whose records will be reviewed in this protocol were enrolled on a number of different protocols between 2013 and 2016.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with metastatic bladder cancer seen between 2013 and 2016 at the NIH Clinical Center.

EXCLUSION CRITERIA:

Patients who opted out of storage of specimens/data for future use on prior studies will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records from patients with metastatic bladder cancer seen between 2013 and 2016 at the NIH Clinical Center. Protocols from which research data originated are 01C0129, 12C0205, 13C0063, and 15C0160.@@@
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Disease burden | 1 year
  Comparison of measure of disease burden by PET/MRI versus traditional CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States